CLINICAL TRIAL: NCT00510146
Title: Efficacy and Safety of Olanzapine in the Treatment of Patients With Bipolar I Disorder, Depressed: A Randomized, Double-Blind Comparison With Placebo
Brief Title: Olanzapine Treatment of Patients With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11218; F1D-MC-HGMP (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Results first posted 2011-05-26 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-04

CONDITIONS: Depression, Bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Olanzapine (Experimental): During double-blind treatment, participants receive olanzapine at a dose of 5 milligram (mg) which is increased to 10 mg per day no later than 3-7 days after randomization (Baseline). Subsequent dose increases above 10 mg (up to a maximum of 20 mg per day) are permitted in 5 mg per day increments, based upon tolerability and symptoms. Dosing may be decreased by any number of decrements, however dosing below 5 mg requires study discontinuation.
  Interventions: Drug: Olanzapine
- Placebo (Placebo Comparator): Matching placebo administered once daily, by mouth during double-blind treatment.
  Interventions: Drug: Placebo
- Olanzapine (open-label treatment period) (Experimental): During open-label treatment, participants randomized to placebo in double-blind period will receive olanzapine 5 mg starting at Week 6. Participants randomized to olanzapine must be at a 5 mg olanzapine dose at Week 7. Those on higher doses will be reduced between Week 6 and Week 7 (10 mg reduced to 5 mg; 15 mg reduced to 10 mg and then to 5 mg at Week 7; 20 mg reduced to 15 mg and then 10 mg to dosing at 5 mg at Week 7). Dose increases beyond Week 7 are permitted and at the investigator's discretion.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — 5-20 mg, oral, once daily, for 24 weeks (participants randomized to olanzapine in double-blind treatment period) or 18 weeks (participants randomized to placebo in double-blind treatment period).
  Other Names: LY170053; Zyprexa
  Arms: Olanzapine; Olanzapine (open-label treatment period)
Drug: Placebo — placebo tablets, oral, once daily at bedtime, 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether olanzapine is superior to placebo in patients with bipolar depression.

DETAILED DESCRIPTION:
1. Dose range and administration mode: Oral Olanzapine 5mg - 20mg/day
2. Duration:

   1. Screening phase is 2-28 days.
   2. Double-blind treatment phase is 6 weeks
   3. Open-label extension phase is 18 weeks

ELIGIBILITY:
Inclusion Criteria:

* Each patient must be reliable, have a level of understanding sufficient to perform all tests and examinations required by the protocol, and must understand the nature of the study and have provided informed consent
* All female patients must test negative for pregnancy and females of breast-feeding potential must agree not to breastfeed an infant during the study and for 1 month following the last dose of study drug
* Patients must fulfill the criteria for a major depressive episode according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV-TR) as well as criteria for bipolar I disorder, depressed, as defined in the DSM-IV-TR, based on clinical assessment and confirmed by the structured diagnostic interview, the Mini International Neuropsychiatric Interview (MINI), at study entry
* Patients must have a current 17-item Hamilton Depression Rating Scale (HAMD-17) score greater than or equal to 18 at Visit 1 and Visit 2
* Patients must have a current Young Mania Rating Scale (YMRS) total score less than or equal to 8 at Visit 2.

Exclusion Criteria:

* Has received treatment within the past 30 days with a drug (not including study drug) that has not received regulatory approval for any indication at the time of study entry
* Has participated in a clinical trial of another investigational drug, including olanzapine, within 1 month (30 days) before study entry
* Was previously treated with olanzapine and had bipolar depression considered to be treatment-resistant to olanzapine or to olanzapine in combination with an available selective serotonin reuptake inhibitor (SSRI)
* Is experiencing (at the time of study entry) a current episode of bipolar depression that is greater than 90 days in duration
* Has been treatment-resistant to any therapy prescribed for bipolar depression when olanzapine alone or with an SSRI prescribed at an appropriate dose and duration

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 514 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5hrs, EST), Study Director — Eli Lilly and Company
Locations (16):
- China (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harbin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kunming
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an
- Japan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shiga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul

REFERENCES:
- [Derived] Katagiri H, Tohen M, McDonnell DP, Fujikoshi S, Case M, Kanba S, Takahashi M, Gomez JC. Safety and efficacy of olanzapine in the long-term treatment of Japanese patients with bipolar I disorder, depression: an integrated analysis. Psychiatry Clin Neurosci. 2014 Jul;68(7):498-505. doi: 10.1111/pcn.12156. Epub 2014 Mar 4. PMID 24417745
- [Derived] Katagiri H, Tohen M, McDonnell DP, Fujikoshi S, Case M, Kanba S, Takahashi M, Gomez JC. Efficacy and safety of olanzapine for treatment of patients with bipolar depression: Japanese subpopulation analysis of a randomized, double-blind, placebo-controlled study. BMC Psychiatry. 2013 May 14;13:138. doi: 10.1186/1471-244X-13-138. PMID 23672672
- [Derived] Tohen M, McDonnell DP, Case M, Kanba S, Ha K, Fang YR, Katagiri H, Gomez JC. Randomised, double-blind, placebo-controlled study of olanzapine in patients with bipolar I depression. Br J Psychiatry. 2012 Nov;201(5):376-82. doi: 10.1192/bjp.bp.112.108357. Epub 2012 Aug 23. PMID 22918966

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period I (2-28 days) included screening and lead-in period for discontinuation of excluded medications at least 25 hours before day of randomization. Study Period II was 6-week, double-blind (Acute Phase) of treatment. Study Period III was 18-week, open-label extension for those who completed Study Period II.
Groups:
- Olanzapine: During double-blind treatment, participants receive olanzapine at a dose of 5 mg which is increased to 10 mg per day no later than 3-7 days after randomization (Baseline). Subsequent dose increases above 10 mg (up to a maximum of 20 mg per day) are permitted in 5 mg per day increments, based upon tolerability and symptoms. Dosing may be decreased by any number of decrements, however dosing below 5 mg requires study discontinuation.
Period: Double-Blind Treatment
Arm/Group | Olanzapine | Placebo
Started | 343 | 171
Completed | 267 | 122
Not Completed | 76 | 49
Not completed — Adverse Event | 30 | 13
Not completed — Lack of Efficacy | 6 | 13
Not completed — Lost to Follow-up | 3 | 7
Not completed — Physician Decision | 6 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 27 | 13
Not completed — Clinical Relapse | 0 | 1
Not completed — Entry Criteria Not Met | 3 | 0
Period: Open-Label Treatment
Arm/Group | Olanzapine | Placebo
Started | 267 | 122
Completed | 196 | 96
Not Completed | 71 | 26
Not completed — Adverse Event | 22 | 8
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 4 | 0
Not completed — Lost to Follow-up | 10 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 24 | 12
Not completed — Clinical Relapse | 1 | 1
Not completed — Sponsor Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Placebo | Total
Number analyzed (Participants) | 343 | 171 | 514
Age Continuous [Mean (Standard Deviation); unit: years] | 35.93 (11.13) | 34.96 (11.02) | 35.61 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 95 | 300
  Male | 138 | 76 | 214
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 36 | 22 | 58
  African | 18 | 4 | 22
  Hispanic | 6 | 3 | 9
  East Asian | 282 | 141 | 423
  Native American | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  China | 140 | 70 | 210
  Japan | 104 | 52 | 156
  Korea, Republic of | 20 | 10 | 30
  Taiwan | 19 | 9 | 28
  United States | 60 | 30 | 90
Age at onset, Bipolar I Disorder [Mean (Standard Deviation); unit: years] | 27.57 (10.98) | 26.12 (9.90) | 27.09 (10.64)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score (Acute Phase)
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline, Endpoint (Week 6)
Population: Intention-to-treat population (ITT) with non-missing baseline value and at least one non-missing post baseline value, last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 339 | 169
units on a scale
  Baseline | 29.36 (5.71) | 28.69 (6.33)
  Change | -14.26 (9.73) | -11.71 (11.09)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.018, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in MADRS total score from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-3.93 to -0.36]

2. Secondary Outcome: Percentage of Participants With Symptomatic Response at Endpoint (Acute Phase)
Description: Response is defined as a reduction (from baseline to endpoint) of 50% or more in the MADRS total score. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Endpoint (Week 6)
Population: Intention-to-treat (ITT) population; all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 343 | 171
percentage of participants | 52.5 | 43.3
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.050, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with symptomatic response at endpoint from a Cochran-Mantel-Haenszel test using geographic region as strata

3. Secondary Outcome: Percentage of Participants With Symptomatic Remission At Any Time (Acute Phase)
Description: Percentage of participants with symptomatic remission at any time as defined as a score of less than or equal to 12 in the MADRS total score. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline through Endpoint (Week 6)
Population: Intention-to-treat (ITT) population; all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 343 | 171
percentage of participants | 53.9 | 49.7
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.367, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with symptomatic remission at any time from a Cochran-Mantel-Haenszel test using region as strata

4. Secondary Outcome: Change From Baseline to Endpoint in Clinical Global Improvement- Bipolar (CGI-BP) Severity of Illness Scores-Mania, Depression, Overall Bipolar Illness Scores (Acute Phase)
Description: CGI-BP is a measure of illness severity especially adapted for bipolar illness. It allows rating of mania, depression, and overall illness. The score ranges from 1 (normal, not ill) to 7 (very seriously ill).
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 339 | 169
units on a scale
  Baseline-Mania | 1.07 (0.29) | 1.11 (0.35)
  Change-Mania | 0.00 (0.43) | 0.09 (0.59)
  Baseline-Depression | 4.54 (0.73) | 4.53 (0.73)
  Change-Depression | -1.45 (1.26) | -1.20 (1.36)
  Baseline- Overall | 4.45 (0.79) | 4.44 (0.79)
  Change- Overall | -1.40 (1.28) | -1.08 (1.27)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.008, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in CGI-BP Mania score from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region; Median Difference (Final Values) = -0.11, 95% CI 2-sided [-0.20 to -0.03]
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.037, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in CGI-BP Depression score from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region; Median Difference (Final Values) = -0.24, 95% CI 2-sided [-0.47 to -0.01]
Statistical Analysis 3: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.008, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in CGI-BP Overall score from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region; Median Difference (Final Values) = -0.30, 95% CI 2-sided [-0.53 to -0.08]

5. Secondary Outcome: Percentage of Participants With Recovery (Acute Phase)
Description: Percentage of participants with recovery defined as a value of less than or equal to 12 in the MADRS total score for at least 4 weeks of post-baseline treatment. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline through Endpoint (Week 6 )
Population: Intention-to-treat (ITT) population; all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 343 | 171
percentage of participants | 13.7 | 9.4
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.156, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with recovery from a Cochran-Mantel-Haenszel test using region as strata

6. Secondary Outcome: Change From Baseline to Endpoint in Young Mania Rating Scale (YMRS) Total Score (Acute Phase)
Description: The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 339 | 169
units on a scale
  Baseline | 2.14 (2.10) | 1.95 (2.18)
  Change | -0.78 (2.56) | 0.31 (4.21)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-1.56 to -0.43]

7. Secondary Outcome: Change From Baseline to Endpoint in Hamilton Depression Rating Scale-17 (HAMD-17) Total Score (Acute Phase)
Description: The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 318 | 155
units on a scale
  Baseline | 22.62 (3.47) | 22.35 (3.53)
  Change | -11.44 (7.02) | -9.12 (7.99)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -2.21, 95% CI 2-sided [-3.61 to -0.81]

8. Secondary Outcome: Percentage of Participants With Major Depressive Episode at Endpoint on Mini International Neuropsychiatric Interview (MINI), Depressive Episode Module (Acute Phase)
Description: In the MINI Major Depressive Episode module, participants are asked a series of Yes/No questions to determine whether or not they are experiencing a major depressive episode or a major depressive episode with melancholic features.
Time Frame: Endpoint (Week 6)
Population: Intention-to-treat (ITT) population with non-missing baseline value and at least one non-missing post baseline value, last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 339 | 169
percentage of participants
  Major Depressive Episode | 55.5 | 60.4
  Major Depressive Episode with Melancholic Features | 77.8 | 74.1
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.297, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with major depressive episode from a Cochran-Mantel-Haenszel test using geographic region as strata
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.264, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with major depressive episode with melancholic features from a Cochran-Mantel-Haenszel test using geographic region as strata

9. Secondary Outcome: Percentage of Participants With Current Hypomanic Episode at Endpoint on MINI Manic Episode Module (Acute Phase)
Description: In the MINI Manic Episode module, participants are asked a series of Yes/No questions to determine whether or not they are currently experiencing hypomanic or manic episodes.
Time Frame: Endpoint (Week 6)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 332 | 169
percentage of participants | 2.1 | 0.6
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.195, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with current hypomanic episode from a Cochran-Mantel-Haenszel test using geographic region as strata

10. Secondary Outcome: Percentage of Participants With Psychotic Disorders and Mood Disorders With Psychotic Features at Endpoint on MINI Psychotic Disorders Module (Acute Phase)
Description: In the MINI Psychotic Features Episode module, participants are asked a series of Yes/No questions to determine whether or not they are currently experiencing mood disorder with psychotic features or current psychotic disorders.
Time Frame: Endpoint (Week 6)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 339 | 169
percentage of participants
  Mood Disorder with Psychotic Features | 3.6 | 2.4
  Psychotic Disorders | 0.0 | 0.6
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.163, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with current psychotic disorders from a Cochran-Mantel-Haenszel test using geographic region as strata
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.442, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with current mood disorders with psychotic features from a Cochran-Mantel-Haenszel test using geographic region as strata

11. Secondary Outcome: Percentage of Participants With Alcohol Dependence and Abuse at Endpoint on MINI Alcohol Dependence/Abuse Module (Acute Phase)
Description: In the MINI Alcohol Abuse and Dependence Module, participants are asked a series of Yes/No questions to determine whether or not they are currently experiencing symptoms indicating current alcohol dependence or abuse.
Time Frame: Endpoint (Week 6)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 335 | 169
percentage of participants
  Dependence | 0.6 | 0.6
  Abuse | 0.6 | 0.0
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 1.00, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with current alcohol dependence from a Cochran-Mantel-Haenszel test using geographic region as strata
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.324, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with current alcohol abuse from a Cochran-Mantel-Haenszel test using geographic region as strata

12. Secondary Outcome: Percentage of Participants With Non-Alcohol Psychoactive Substance Use Disorder at Endpoint on MINI Substance Dependence/Abuse Module (Acute Phase)
Description: In the MINI Substance Dependence and Abuse Module, participants are asked a series of Yes/No questions to determine whether or not they are currently experiencing symptoms indicating current non-alcohol substance use dependence or abuse.
Time Frame: Endpoint (Week 6)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 335 | 169
percentage of participants
  Dependence | 0.0 | 0.0
  Abuse | 0.0 | 0.0

13. Secondary Outcome: Percentage of Participants With Emergence of Mania During the Study (Acute Phase)
Description: Emergence of mania is defined as first occurrence of score of >=15 in the YMRS total score in the post-baseline period of Acute Phase. The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
Time Frame: Baseline through Endpoint (Week 6)
Population: Intention-to-treat (ITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 343 | 171
percentage of participants | 0.6 | 2.9
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.031, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with emergence of mania at endpoint from a Cochran-Mantel-Haenszel test using geographic region as strata

14. Secondary Outcome: Percentage of Participants With Extra-Pyramidal Symptoms (EPS) At Endpoint As Measured by Drug-Induced Extra-Pyramidal Symptoms Scale (DIEPSS) (Acute Phase)
Description: EPS symptoms measured by DIEPSS are grouped into 4 categories: parkinsonism, akathisia, dystonia, and dyskinesia. Severity is assessed at 5 levels, from level 0 (none, normal) to level 4 (severe). For Parkinsonism, normal baseline is defined as a score not >=3 on 1 item nor >=2 on 2 items; abnormal endpoint is defined as a score >=3 on 1 item or >=2 on 2 items, or an increase of 3 on Parkinsonism total. Baseline akathisia, dystonia and dyskinesia is defined as a score <2; abnormal endpoint is a score >=2 or an increase >= 2 from that baseline score.
Time Frame: Endpoint (Week 6)
Population: Participants with a normal baseline and an endpoint result.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 337 | 169
percentage of participants
  Akathisia (N=335, 169) | 2.7 | 1.2
  Dyskinesia (N=337, 169) | 0.0 | 0.0
  Dystonia (N=337, 169) | 0.0 | 0.0
  Parkinsonism (N=337, 169) | 0.9 | 0.6
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.269, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with EPS symptoms (akathisia) at endpoint from a Cochran-Mantel-Haenszel test using geographic region as strata
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.736, Cochran-Mantel-Haenszel — p-value represents a comparison of the olanzapine and placebo groups in percentage of participants with EPS symptoms (parkinsonism) at endpoint from a Cochran-Mantel-Haenszel test using geographic region as strata

15. Secondary Outcome: Change From Baseline to Endpoint in Blood Pressure (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: Safety population; participants with non-missing baseline value and at least one non-missing post baseline value, last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: mmHg (millimeters of mercury)
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 320 | 159
mmHg (millimeters of mercury)
  Baseline- Standing Systolic (N=320, 159) | 112.39 (13.25) | 115.65 (14.39)
  Change- Standing Systolic (N=320, 159) | -0.99 (10.83) | -0.67 (11.18)
  Baseline- Sitting Systolic (N=340, 169) | 112.35 (13.42) | 114.39 (13.67)
  Change- Sitting Systolic (N=340, 169) | -0.36 (11.10) | 0.04 (12.16)
  Baseline- Standing Diastolic (N=320, 159) | 74.77 (10.20) | 76.87 (10.26)
  Change- Standing Diastolic (N=320, 159) | -0.48 (8.71) | -0.14 (8.44)
  Baseline- Sitting Diastolic (N=340, 169) | 73.07 (9.93) | 73.92 (9.86)
  Change- Sitting Diastolic (N=340, 169) | -0.11 (9.37) | 0.39 (9.08)
  Baseline- Orthostatic Change-Systolic (N=320, 159) | 0.54 (6.51) | 1.21 (7.67)
  Change- Orthostatic Change-Systolic (N=320, 159) | -0.65 (8.20) | -0.45 (11.45)
  Baseline- Orthostatic Change-Diastolic (N=320, 159 | 1.92 (5.93) | 2.96 (5.57)
  Change- Orthostatic Change-Diastolic (N=320, 159) | -0.52 (6.79) | -0.47 (6.78)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.146, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-standing systolic blood pressure from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.249, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-sitting systolic blood pressure from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region
Statistical Analysis 3: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.146, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-standing diastolic blood pressure from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region
Statistical Analysis 4: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.271, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-sitting diastolic blood pressure from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region
Statistical Analysis 5: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.284, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-orthostatic change in systolic blood pressure from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region
Statistical Analysis 6: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.067, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-orthostatic change in diastolic blood pressure from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region

16. Secondary Outcome: Change From Baseline to Endpoint in Weight (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 340 | 169
kilograms
  Baseline | 66.11 (18.11) | 68.30 (18.73)
  Endpoint | 2.45 (2.82) | -0.13 (2.10)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-in weight from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region

17. Secondary Outcome: Change From Baseline to Endpoint in Glucose and Lipids (Cholesterol, Triglycerides, HDL Cholesterol, LDL Cholesterol)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 329 | 160
millimole/Liter
  Baseline- Fasting Glucose (N=320, 155) | 5.11 (0.58) | 5.12 (0.57)
  Change- Fasting Glucose (N=320, 155) | 0.10 (0.61) | 0.02 (0.54)
  Baseline- Cholesterol (N=329, 160) | 4.83 (1.01) | 4.81 (1.00)
  Change- Cholesterol (N=329, 160) | 0.24 (0.76) | -0.07 (0.49)
  Baseline-Triglycerides (N=329, 160) | 1.39 (0.85) | 1.34 (0.80)
  Change- Triglycerides (N=329, 160) | 0.26 (0.97) | 0.03 (0.71)
  Baseline- LDL Cholesterol (N=328, 159) | 2.77 (0.87) | 2.83 (0.84)
  Change- LDL Cholesterol (N=328, 159) | 0.17 (0.66) | -0.09 (0.48)
  Baseline- HDL Cholesterol (N=329, 160) | 1.43 (0.41) | 1.36 (0.35)
  Change- HDL Cholesterol (N=329, 160) | -0.03 (0.25) | 0.02 (0.21)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.179, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-in fasting glucose from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-in cholesterol from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region
Statistical Analysis 3: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-in triglycerides from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region
Statistical Analysis 4: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-in LDL cholesterol from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region
Statistical Analysis 5: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.095, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint-in HDL cholesterol from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region

18. Secondary Outcome: Change From Baseline to Endpoint in Albumin (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: gram/Liter
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 329 | 160
gram/Liter
  Baseline | 43.07 (3.85) | 43.47 (3.69)
  Change | -0.81 (2.89) | 0.03 (3.11)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in albumin from Wilcoxon's rank-sum test

19. Secondary Outcome: Change From Baseline to Endpoint in Alanine Amino Transferase/Serum Glutamate Pyruvate Transaminase (ALT/SGPT), Aspartate Aminotransferase/Serum Glutamic Oxaloacetic Transaminase (AST/SGOT), Gamma Glutamyl Transferase (GGT)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units/Liter
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 329 | 160
units/Liter
  Baseline (ALT/SGPT) | 21.68 (16.53) | 21.18 (13.17)
  Change (ALT/SGPT) | 8.34 (26.90) | 0.00 (13.63)
  Baseline (AST/SGOT) | 21.61 (8.34) | 20.25 (6.70)
  Change (AST/SGOT) | 4.31 (15.66) | 1.26 (11.06)
  Baseline (GGT) | 24.87 (36.59) | 23.63 (23.17)
  Change (GGT) | 5.36 (22.70) | -1.21 (11.67)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in ALT/SGPT from Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in AST/SGOT from Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in GGT from Wilcoxon's rank-sum test

20. Secondary Outcome: Change From Baseline to Endpoint in Direct Bilirubin, Total Bilirubin, Uric Acid (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 329 | 160
micromole/Liter
  Baseline- Direct Bilirubin | 2.45 (1.23) | 2.40 (1.08)
  Change- Direct Bilirubin | -0.21 (1.03) | 0.12 (1.02)
  Baseline- Total Bilirubin | 9.74 (5.18) | 9.42 (4.58)
  Change- Total Bilirubin | -0.68 (4.57) | 0.47 (4.27)
  Baseline- Uric Acid | 307.19 (92.03) | 314.38 (86.69)
  Change- Uric Acid | 19.55 (51.10) | -1.86 (50.37)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in direct bilirubin from Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in total bilirubin from Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in uric acid from Wilcoxon's rank-sum test

21. Secondary Outcome: Change From Baseline to Endpoint in Erythrocyte Count (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: trillion cells per liter ( TRIL/L)
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 328 | 158
trillion cells per liter ( TRIL/L)
  Baseline | 4.65 (0.51) | 4.71 (0.52)
  Change | -0.05 (0.27) | 0.02 (0.27)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in erythrocyte count from Wilcoxon's rank-sum test

22. Secondary Outcome: Change From Baseline to Endpoint in Hematocrit (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: proportion of blood volume
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 328 | 158
proportion of blood volume
  Baseline | 0.42 (0.04) | 0.43 (0.05)
  Change | -0.01 (0.03) | 0.00 (0.03)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in hematocrit from Wilcoxon's rank-sum test

23. Secondary Outcome: Change From Baseline to Endpoint in Hemoglobin A1c (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent of glycosylated hemoglobin
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 312 | 146
percent of glycosylated hemoglobin
  Baseline | 5.34 (0.37) | 5.37 (0.37)
  Change | 0.04 (0.26) | -0.03 (0.28)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.009, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in hemoglobin A1c from Wilcoxon's rank-sum test

24. Secondary Outcome: Change From Baseline to Endpoint in Hemoglobin (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: millimole/Liter of iron (Fe)
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 328 | 158
millimole/Liter of iron (Fe)
  Baseline | 8.65 (0.99) | 8.73 (0.97)
  Change | -0.11 (0.50) | 0.05 (0.50)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in hemoglobin from Wilcoxon's rank-sum test

25. Secondary Outcome: Change From Baseline to Endpoint in Prolactin (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: microgram/Liter
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 318 | 147
microgram/Liter
  Baseline | 15.40 (16.89) | 15.86 (21.54)
  Change | 12.07 (24.00) | -1.18 (26.49)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in prolactin from Wilcoxon's rank-sum test

26. Secondary Outcome: Change From Baseline to Endpoint in Urinalysis (UA)- Specific Gravity (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 314 | 148
ratio
  Baseline | 1.02 (0.01) | 1.02 (0.01)
  Change | -0.00 (0.01) | 0.00 (0.01)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in urinalysis-specific gravity from Wilcoxon's rank-sum test

27. Secondary Outcome: Change in Electrocardiogram (ECG) From Baseline to Endpoint (Acute Phase)
Description: Time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole, fixed correction factor (QTcF interval); Bazett-Corrected QT Interval (QTcB interval).
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 295 | 145
milliseconds
  Baseline- QTcF | 406.85 (19.53) | 408.10 (18.72)
  Change- QTcF | 2.82 (14.21) | 0.50 (12.27)
  Baseline- QTcB | 415.79 (20.55) | 418.42 (19.95)
  Change- QTcB | 6.58 (18.01) | 1.21 (16.02)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.104, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in QTcF interval from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.006, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in QTcB interval from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region

28. Secondary Outcome: Change From Baseline to Endpoint in Heart Rate (Acute Phase)
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 309 | 148
beats per minute (bpm)
  Baseline | 69.63 (12.65) | 70.51 (11.94)
  Change | 3.49 (11.18) | 0.87 (11.51)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.035, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint in heart rate from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region

29. Secondary Outcome: Change From Baseline to Endpoint in MINI Suicidality Total Scores (Acute Phase)
Description: The MINI module C (MINI-C) is a rating scale for severity of suicidal thoughts and behaviors. The MINI-C is composed of 12 Yes/No questions with variable scores assigned to each question. The scale ranges from 0 to 52 with higher scores indicating a greater presence of suicidal thoughts and/or behaviors.
Time Frame: Baseline, Endpoint (Week 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 337 | 169
units on a scale
  Baseline | 2.09 (3.44) | 2.40 (3.49)
  Change | -0.42 (3.71) | -0.59 (3.44)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.943, ANCOVA — p-value represents a comparison of the olanzapine and placebo groups in change from baseline to endpoint for MINI Suicidality Total Score from the following ANCOVA model: Change=Treatment+Baseline+Geographic Region; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.59 to 0.64]

30. Secondary Outcome: Number of Participants With Adverse Events (Acute Phase)
Description: Please refer to the Adverse Event overview for details regarding adverse events and serious adverse events.
Time Frame: Baseline through Week 6 (Acute Phase)
Population: All enrolled participants in Acute Phase
Measure: Number; unit: participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 343 | 171
participants
  Serious | 6 | 7
  Non-Serious | 238 | 88

31. Secondary Outcome: Percentage of Participants With Symptomatic Response in Montgomery-Asberg Depression Rating (MADRS) Depression Rating (Open-Label Phase)
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Response is defined as a reduction (from baseline to endpoint) of 50% or more in the MADRS total score.
Time Frame: Baseline (End of Acute Phase/Week 6) through Endpoint (Week 24)
Population: Total participants in the open-label extension phase.
Measure: Number; unit: percentage of participants
Groups:
- Olanzapine (Open-label Treatment Period): During open-label treatment, participants randomized to placebo in double-blind period will receive olanzapine 5 mg starting at Week 6. Participants randomized to olanzapine must be at a 5 mg olanzapine dose at Week 7. Those on higher doses will be reduced between Week 6 and 7 (10 mg reduced to 5 mg; 15 mg reduced to 10 mg and then to 5 mg at Week 7; 20 mg reduced to 15 mg and then 10 mg to dosing at 5 mg at Week 7). Dose increases beyond Week 7 are permitted and at the investigator's discretion.
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 389
percentage of participants | 43.7

32. Secondary Outcome: Percentage of Participants With Symptomatic Remission in the MADRS Total Score (Open-Label Phase)
Description: as for outcome 3
Time Frame: Baseline (End of Acute Phase/Week 6) through Endpoint (Week 24)
Population: Total participants in open-label extension phase.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 389
percentage of participants | 85.1

33. Secondary Outcome: Percentage of Participants With Recovery (Open-Label Phase)
Description: as for outcome 5
Time Frame: Baseline (End of Acute Phase/Week 6) through Endpoint (Week 24)
Population: Total participants in open-label extension phase.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 389
percentage of participants | 69.9

34. Secondary Outcome: Change From Baseline to Endpoint in Young Mania Rating Scale (YMRS) Total Score (Open-Label Phase)
Description: as for outcome 6
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: Participants who entered Open-Label Phase with non-missing baseline (end of Acute Phase) and post-baseline visit, last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 385
units on a scale
  Baseline | 1.11 (2.87)
  Change | -0.03 (2.55)

35. Secondary Outcome: Percentage of Participants With Emergence of Mania During the Study (Open-Label Phase)
Description: Emergence of mania is defined as first occurrence of score of >=15 in the YMRS total score in the Open-Label Extension. The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
Time Frame: Baseline (End of Acute Phase/Week 6) through Endpoint (Week 24)
Population: Total participants in the open-label extension phase.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 389
percentage of participants | 0.8

36. Secondary Outcome: Percentage of Participants With Extra-Pyramidal Symptoms (EPS) at Endpoint As Measured by Drug-Induced Extra-Pyramidal Symptoms Scale (DIEPSS) (Open-Label Phase)
Description: as for outcome 14
Time Frame: Endpoint (Week 24)
Population: Participants who entered Open-Label Phase with a normal baseline and at least one post-baseline result.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 385
percentage of participants
  Akathisia (N=378) | 0.8
  Dyskinesia (N=385) | 0.3
  Dystonia (N=385) | 0.0
  Parkinsonism (N=385) | 1.0

37. Secondary Outcome: Change From Baseline to Endpoint in Blood Pressure (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 383
millimeters of mercury
  Baseline-Standing Diastolic (N=361) | 74.98 (10.77)
  Change- Standing Diastolic (N=361) | 0.15 (8.28)
  Baseline- Sitting Diastolic (N=383) | 73.32 (10.73)
  Change- Sitting Diastolic (N=383) | -0.03 (8.68)
  Baseline- Standing Systolic (N=361) | 112.06 (14.58)
  Change- Standing Systolic (N=361) | 0.96 (10.37)
  Baseline- Sitting Systolic (N=383) | 112.26 (14.45)
  Change- Sitting Systolic (N=383) | 0.27 (10.28)
  Baseline- Orthostatic Change-Diastolic (N=358) | 1.75 (5.25)
  Change- Orthostatic Change- Diastolic (N=358) | 0.16 (6.56)
  Baseline- Orthostatic Change- Systolic (N=358) | 0.19 (6.19)
  Change- Orthostatic Change- Systolic (N=358) | 0.65 (7.92)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.736, t-test, 2 sided — p-value represents change from baseline to endpoint-standing diastolic blood pressure from t-tests on change
Statistical Analysis 2: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.944, t-test, 2 sided — p-value represents change from baseline to endpoint-sitting diastolic blood pressure from t-tests on change
Statistical Analysis 3: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.080, t-test, 2 sided — p-value represents change from baseline to endpoint-standing systolic blood pressure from t-tests on change
Statistical Analysis 4: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.612, t-test, 2 sided — p-value represents change from baseline to endpoint-sitting systolic blood pressure from t-tests on change
Statistical Analysis 5: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.640, t-test, 2 sided — p-value represents change from baseline to endpoint-orthostatic change in diastolic blood pressure from t-tests on change
Statistical Analysis 6: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.122, t-test, 2 sided — p-value represents change from baseline to endpoint-orthostatic change in systolic blood pressure from t-tests on change

38. Secondary Outcome: Change From Baseline to Endpoint in Weight (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/ Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 384
kilograms
  Baseline | 68.31 (18.54)
  Change | 2.27 (4.00)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value represents change from baseline to endpoint for weight from t-tests on change

39. Secondary Outcome: Change From Baseline to Endpoint in Albumin and Total Protein (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: gram/Liter
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 381
gram/Liter
  Baseline- Albumin | 42.64 (3.58)
  Change- Albumin | 0.53 (2.86)
  Baseline- Total Protein | 73.24 (4.39)
  Change- Total Protein | 0.56 (3.78)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for albumin from Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for total protein from Wilcoxon's signed-rank test

40. Secondary Outcome: Change From Baseline to Endpoint in Alkaline Phosphatase, Creatinine Phosphokinase (CPK), GGT (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: units/Liter
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 381
units/Liter
  Baseline- Alkaline Phosphatase | 68.58 (19.33)
  Change- Alkaline Phosphatase | 2.37 (12.85)
  Baseline- CPK | 107.36 (133.21)
  Change- CPK | -1.73 (124.56)
  Baseline- GGT | 28.90 (32.08)
  Change- GGT | 0.78 (25.90)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for alkaline phosphatase from Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for CPK from Wilcoxon's signed-rank test
Statistical Analysis 3: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.354, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for GGT from Wilcoxon's signed-rank test

41. Secondary Outcome: Change From Baseline to Endpoint in Chloride (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 381
millimole/Liter
  Baseline | 103.62 (2.16)
  Change | 0.33 (2.38)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for chlorine from Wilcoxon's signed-rank test

42. Secondary Outcome: Change From Baseline to Endpoint in Creatinine (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 381
micromole/Liter
  Baseline | 67.48 (14.98)
  Change | 2.05 (7.90)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for creatinine from Wilcoxon's signed-rank test

43. Secondary Outcome: Change From Baseline to Endpoint in Erythrocyte Count (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: trillion cells per liter (Tril/L)
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 380
trillion cells per liter (Tril/L)
  Baseline | 4.64 (0.53)
  Change | 0.03 (0.30)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.021, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for erythrocyte count from Wilcoxon's signed-rank test

44. Secondary Outcome: Change From Baseline to Endpoint in Hemoglobin (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: millimole/Liter of iron (Fe)
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 380
millimole/Liter of iron (Fe)
  Baseline | 8.61 (1.01)
  Change | 0.04 (0.51)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.035, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for hemoglobin from Wilcoxon's signed-rank test

45. Secondary Outcome: Change From Baseline to Endpoint in Platelet Count (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: billion cells per liter (BILL/L)
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 380
billion cells per liter (BILL/L)
  Baseline | 257.96 (64.25)
  Change | -4.56 (49.94)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.024, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for platelet count from Wilcoxon's signed-rank test

46. Secondary Outcome: Change From Baseline to Endpoint in Prolactin (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: microgram/Liter
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 346
microgram/Liter
  Baseline | 21.64 (18.48)
  Change | -3.41 (17.20)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for prolactin from Wilcoxon's signed-rank test

47. Secondary Outcome: Change From Baseline to Endpoint in Uric Acid (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 381
micromole/Liter
  Baseline | 324.74 (89.39)
  Change | 14.73 (56.80)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — p-value represents change from baseline to endpoint for uric acid from Wilcoxon's signed-rank test

48. Secondary Outcome: Change From Baseline to Endpoint in Glucose and Lipids (Cholesterol, Triglycerides, HDL Cholesterol, LDL Cholesterol) (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 380
millimole/Liter
  Baseline- Fasting Glucose (N=375) | 5.20 (0.57)
  Change- Fasting Glucose (N=375) | 0.06 (0.63)
  Baseline- Cholesterol (N=380) | 4.96 (1.08)
  Change- Cholesterol (N=380) | 0.05 (0.70)
  Baseline- Triglycerides (N=380) | 1.55 (1.06)
  Change- Triglycerides (N=380) | 0.10 (0.97)
  Baseline- LDL Cholesterol (N=378) | 2.88 (0.91)
  Change- LDL Cholesterol (N=378) | 0.06 (0.63)
  Baseline- HDL Cholesterol (N=380) | 1.39 (0.40)
  Change- HDL Cholesterol (N=380) | -0.05 (0.24)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.047, t-test, 2 sided — p-value represents change from baseline to endpoint for fasting glucose from t-tests on change
Statistical Analysis 2: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.130, t-test, 2 sided — p-value represents change from baseline to endpoint for cholesterol from t-tests on change
Statistical Analysis 3: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.055, t-test, 2 sided — p-value represents change from baseline to endpoint for triglycerides from t-tests on change
Statistical Analysis 4: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.049, t-test, 2 sided — p-value represents change from baseline to endpoint for LDL cholesterol from t-tests on change
Statistical Analysis 5: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value represents change from baseline to endpoint for HDL cholesterol from t-tests on change

49. Secondary Outcome: Change From Baseline to Endpoint in ECG (Open-Label Phase)
Description: as for outcome 27
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 366
milliseconds
  Baseline- QTcF | 410.09 (19.44)
  Change- QTcF | 1.80 (15.07)
  Baseline- QTcB | 421.72 (19.61)
  Change- QTcB | 1.76 (16.69)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.023, t-test, 2 sided — p-value represents change from baseline to endpoint for QTcF from t-test
Statistical Analysis 2: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.044, t-test, 2 sided — p-value represents change from baseline to endpoint for QTcB from t-test

50. Secondary Outcome: Change From Baseline to Endpoint in Heart Rate (Open-Label Phase)
Time Frame: Baseline (End of Acute Phase/Week 6), Endpoint (Week 24)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 370
beats per minute
  Baseline | 71.85 (11.64)
  Change | 0.06 (10.79)
Statistical Analysis 1: Comparison: Olanzapine (Open-label Treatment Period); Test type: Superiority or Other; p = 0.919, t-test, 2 sided — p-value represents change from baseline to endpoint for heart rate from t-test

51. Secondary Outcome: Percentage of Participants With High Suicidality at Endpoint (Open-Label Phase)
Description: The MINI module C (MINI-C) is a rating scale for severity of suicidal thoughts and behaviors. The MINI-C is composed of 12 Yes/No questions with variable scores assigned to each question. The scale ranges from 0 to 52 with higher scores indicating a greater presence of suicidal thoughts and/or behaviors. Based upon scores, suicidality is defined as Low (1-8), Medium (9-16), and High (>=17).
Time Frame: Endpoint (Week 24)
Population: Total participants in the open-label extension phase.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 389
percentage of participants | 1.3

52. Secondary Outcome: Number of Participants With Adverse Events (Open-Label Phase)
Description: Please refer to the Adverse Event overview for details regarding adverse events and serious adverse events.
Time Frame: Baseline (End of Acute Phase/Week 6) through Endpoint (Week 24)
Population: Total participants in the open-label extension phase.
Measure: Number; unit: participants
Arm/Group | Olanzapine (Open-label Treatment Period)
Number analyzed (Participants) | 389
participants
  Serious | 14
  Non-Serious | 209

ADVERSE EVENTS:
Groups:
- Olanzapine: During double-blind treatment, participants receive olanzapine at a dose of 5 mg. which is increased to 10 mg. per day no later than 3-7 days after Visit 2. Subsequent dose increases above 10 mg. (up to a maximum of 20 mg per day) are permitted in 5 mg. per day increments, based upon tolerability and symptoms. Dosing may be decreased by any number of decrements, however dosing below 5 mg. requires study discontinuation.
- Olanzapine (Open Label Treatment Period: During open-label treatment, participants randomized to placebo in double-blind period will receive olanzapine 5 mg starting at Visit 9. Participants randomized to olanzapine must be at a 5 mg olanzapine dose at Visit 10. Those on higher doses will be reduced between Visit 9 and 10 (10 mg reduced to 5 mg; 15 mg reduced to 10 mg and then to 5 mg at visit 10; 20 mg reduced to 15 mg and then 10 mg to dosing at 5 mg at visit 10). Dose increases beyond visit 10 are permitted and at the investigator's discretion.
Arm/Group | Olanzapine | Placebo | Olanzapine (Open Label Treatment Period
Serious Adverse Events (participants affected / at risk) | 6/343 | 7/171 | 14/389
Other Adverse Events (participants affected / at risk) | 238/343 | 88/171 | 209/389
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=343) | Placebo (N=171) | Olanzapine (Open Label Treatment Period (N=389)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=343) | Placebo (N=171) | Olanzapine (Open Label Treatment Period (N=389)
Constipation (Gastrointestinal disorders) | 19 (21) | 5 (5) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 6 (6) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 18 (18) | 6 (6) | 4 (4)
Nausea (Gastrointestinal disorders) | 7 (7) | 8 (9) | 4 (4)
Fatigue (General disorders) | 10 (10) | 6 (8) | 3 (3)
Thirst (General disorders) | 11 (11) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 11 (11) | 1 (1) | 6 (6)
Nasopharyngitis (Infections and infestations) | 24 (25) | 6 (6) | 20 (25)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 6 (7) | 3 (3)
Alanine aminotransferase increased (Investigations) | 11 (11) | 0 (0) | 12 (13)
Weight increased (Investigations) | 59 (59) | 6 (6) | 67 (67)
Increased appetite (Metabolism and nutrition disorders) | 46 (46) | 4 (5) | 15 (15)
Akathisia (Nervous system disorders) | 14 (14) | 2 (2) | 9 (9)
Dizziness (Nervous system disorders) | 13 (13) | 6 (6) | 6 (6)
Headache (Nervous system disorders) | 15 (17) | 8 (9) | 10 (12)
Hypersomnia (Nervous system disorders) | 15 (15) | 2 (2) | 14 (14)
Sedation (Nervous system disorders) | 29 (33) | 4 (4) | 3 (3)
Somnolence (Nervous system disorders) | 59 (60) | 11 (11) | 17 (20)
Tremor (Nervous system disorders) | 14 (15) | 5 (5) | 7 (7)
Anxiety (Psychiatric disorders) | 11 (13) | 5 (5) | 10 (10)
Insomnia (Psychiatric disorders) | 11 (11) | 8 (8) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days